CLINICAL TRIAL: NCT05963581
Title: Investigating the Effects of Social Movement on Mood and Social and Emotional Functioning in Young People Experiencing Low Mood
Brief Title: Oxford Social Movement Activation Study
Acronym: SOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SOMA
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Depression; Low Mood; Depressive Disorder; Mood Disorders; Depressive Symptoms
Keywords: low mood, depression, social movement, dance, salsa dance
MeSH Terms: conditions — Depression; Consciousness Disorders; Depressive Disorder; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the salsa dancing intervention (46 participants) or the passive waiting-list control group (46 participants). Randomization will be stratified by gender.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salsa Dancing (Experimental): Participants will complete eight weeks of a salsa course in Oxford (of which they need to attend six classes to remain in the study), followed by a one-month follow-up time point.
  Interventions: Behavioral: Salsa Dancing
- Waitlist Control (No Intervention): Participants will wait twelve weeks, completing the questionnaires and tasks at the same study time points as participants in the experimental condition.They will then be offered the opportunity to complete the eight-week salsa course. Should they choose to participate in the salsa course, they will additionally be offered the opportunity to complete questionnaires at two additional time points.

INTERVENTIONS:
Behavioral: Salsa Dancing — Participants will complete salsa dancing classes in central Oxford with instructor(s) from the Oxford University Salsa Society
  Arms: Salsa Dancing

SUMMARY:
For adolescents and young people particularly, there is need for better and more readily available treatments for depression and low mood. Comparatively less work has been done to characterize and treat depression specifically in young people. Previous literature indicates that often the unaddressed or under-addressed mental health difficulties in youth perseverate into adulthood and contribute to a host of individual and communal difficulties throughout the lifespan. Specifically, if depression goes unaddressed in young adulthood, the likelihood of a chronic course and multiple relapses or recurrences is much higher.

In the present research, we seek to investigate the potential efficacy of a novel intervention for young people with low mood. Depression disrupts social functioning, and social connectedness is especially important during adolescence for healthy development. Within a growing body of literature, social dance has been linked to social and mental health benefits along the dimensions of those disrupted in depression. We hypothesize that social dance might preferentially and efficiently target the goals of addressing loneliness, closeness, and enjoyment in young people compared to other approaches to the treatment of low mood and depression in a way that could lead to mood improvements.

Specifically, we are interested in the impact of a social movement-based activity, salsa dancing, on young peoples' mood and social and emotional processing. Social and emotional processing (SEP) tasks, such as emotional facial recognition and memory for emotional words, have been demonstrated to correspond with early changes that can be predictive of mood changes and treatment efficacy downstream. Including SEP tasks in this research will help to elucidate the potential mechanisms underlying mood improvements, should social dance correspond to improved mood in participants.

The present research seeks to:

1. Aim 1: Investigate the effect of a social dance intervention on low mood. This will be assessed by administering psychological questionnaires to participants before, during, and after the study course of social dance sessions. In particular, we hypothesize that participants will experience reductions in low mood (assessed via the PHQ-9) following the social movement intervention as compared to a waitlist control.
2. Aim 2: Characterize any early social and emotional processing changes that correspond to social dance versus a waitlist control. This will be assessed via social and emotional processing task performance before, during, and following the social movement sessions. We anticipate that improvements in social and emotional functioning as demonstrated via one or several of these tasks will assist in elucidating the possible mechanisms responsible for mood improvement from social movement.
3. Aim 3: Characterize any social interaction difference from pre to post intervention that correspond to the social dance versus waitlist condition. This will be assessed via a version of the trust game before and following the social movement sessions and waitlist control. We anticipate seeing more disrupted trust behavior prior to the intervention or control conditions and less disrupted trust behavior following salsa dancing classes, but not the waitlist control.

In this randomized controlled trial, participants in the experimental group will complete six to eight sessions of social movement (salsa dance) classes within an eight-week period, and complete psychological questionnaires and tasks before, during, and after these eight weeks. Their scores will be compared with those of a control group that will participate in an active waitlist condition.

If the present study suggests that social movement benefits young people with low mood, it could form the basis for investigating a potential new cost-effective, non-invasive, accessible intervention that could be made available to young people.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 24 at time of eligibility screening;
* Competency to give informed consent;
* Individuals will *not* be excluded for a formal diagnosis of depression from a GP or other mental healthcare provider, nor for being presently or formerly on medication for depression; nor for presently or formerly attending talk therapies;
* Individuals who do not meet the exclusion criteria specified below.

Exclusion Criteria:

* Individuals with a PHQ-9 score of less than 5 (indicating no low mood) or greater than 19 (indicating a low mood that could be too severe for this research);
* individuals who self-report a current or recent diagnosis of any psychotic disorder (e.g., bipolar, schizophrenia, schizoaffective disorder), substance use disorders, eating disorders, or personality disorders
* individuals who self-report that they are unfit for light physical exertion;
* individuals who regularly, or have regularly, attended partner dance classes or partner dance events within the last six months (as they would already be receiving the potential benefits we are investigating in this study);
* and individuals for whom the Principal Investigator determines that the study is not suitable.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms from baseline at week four, eight, and twelve | Will be assessed at week 0, 4, 8, and 12 of the intervention
  Patient Health Questionnaire (PHQ-9) score. Higher scores indicate greater depressive symptoms.

SECONDARY OUTCOMES:
Change in anxiety symptoms from baseline at week four, eight, and twelve | Will be assessed at week 0, 4, 8, and 12 of the intervention
  Generalized Anxiety Disorder Scale (GAD-7) score. Higher scores indicate greater anxiety.
Change in social anxiety symptoms from baseline at week four, eight, and twelve | Will be assessed at week 0, 4, 8, and 12 of the intervention
  Social Anxiety Scale - Adolescent (SAS-A) score. Higher scores indicate greater social anxiety.
Change in loneliness from baseline at week four, eight, and twelve | Will be assessed at week 0, 4, 8, and 12 of the intervention
  UCLA Loneliness Scale (+ Loneliness Question) score. Higher scores indicate more loneliness.
Change in daily mood questionnaire scores | daily from baseline through week 12 of the intervention
  Scoring one Likert scale mood questionnaire ("How happy do you feel?"), range 1-10. Higher values represent more happiness.
Change in social anhedonia from baseline at week four, eight, and twelve | Will be assessed at week 0, 4, 8, and 12 of the intervention
  Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) score. Higher scores indicate lower social anhedonia.
Change in recognition of positive and negative facial expressions from baseline at week 8 | Will be assessed at week 0 and week 8 of the intervention
  Hit rate for detecting positive versus negative faces in a facial expression recognition task (FERT)
Change in speed during recognition of positive and negative facial expressions | Will be assessed at week 0 and week 8 of the intervention
  Reaction times for correctly recognised positive versus negative faces in facial expression recognition task (FERT)
Change in emotional categorisation (ECAT) | Will be assessed at week 0 and week 8 of the intervention
  Reaction times for correctly classifying positive versus negative personality characteristic words
Change in recall in the emotional recall task (EREC) | Will be assessed at week 0 and week 8 of the intervention
  Number of positive and negative words correctly (and incorrectly) recalled in the EREC task
Change in memory in the emotional memory task (EMEM) | Will be assessed at week 0 and week 8 of the intervention
  Number of positive and negative words correctly (and incorrectly) recalled as familiar and novel
Change in trust behavior in the trust game (Trust Game) | Will be assessed at week 0 and week 8 of the intervention
  Investment behavior and sensitivity to trustee's generosity when playing the role of the investor in a trust game

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saunders R, Buckman JEJ, Stott J, Leibowitz J, Aguirre E, John A, Lewis G, Cape J, Pilling S; NCEL network. Older adults respond better to psychological therapy than working-age adults: evidence from a large sample of mental health service attendees. J Affect Disord. 2021 Nov 1;294:85-93. doi: 10.1016/j.jad.2021.06.084. Epub 2021 Jul 9. PMID 34274792
- [Background] Buckman JEJ, Underwood A, Clarke K, Saunders R, Hollon SD, Fearon P, Pilling S. Risk factors for relapse and recurrence of depression in adults and how they operate: A four-phase systematic review and meta-synthesis. Clin Psychol Rev. 2018 Aug;64:13-38. doi: 10.1016/j.cpr.2018.07.005. Epub 2018 Jul 29. PMID 30075313
- [Background] Lakes KD, Marvin S, Rowley J, Nicolas MS, Arastoo S, Viray L, Orozco A, Jurnak F. Dancer perceptions of the cognitive, social, emotional, and physical benefits of modern styles of partnered dancing. Complement Ther Med. 2016 Jun;26:117-22. doi: 10.1016/j.ctim.2016.03.007. Epub 2016 Mar 9. PMID 27261991
- [Background] Shuper Engelhard E, Vulcan M. The Potential Benefits of Dance Movement Therapy in Improving Couple Relations of Individuals Diagnosed With Autism Spectrum Disorder-A Review. Front Psychol. 2021 Feb 18;12:619936. doi: 10.3389/fpsyg.2021.619936. eCollection 2021. PMID 33679534
- [Background] Hyvonen K, Pylvanainen P, Muotka J, Lappalainen R. The Effects of Dance Movement Therapy in the Treatment of Depression: A Multicenter, Randomized Controlled Trial in Finland. Front Psychol. 2020 Aug 12;11:1687. doi: 10.3389/fpsyg.2020.01687. eCollection 2020. PMID 32903394
- [Background] Harmer CJ, Duman RS, Cowen PJ. How do antidepressants work? New perspectives for refining future treatment approaches. Lancet Psychiatry. 2017 May;4(5):409-418. doi: 10.1016/S2215-0366(17)30015-9. Epub 2017 Jan 31. PMID 28153641